CLINICAL TRIAL: NCT02680509
Title: Single-port Thoracoscopic Sympathicotomy for Treatment of Raynaud's Phenomenon, a Feasibility Study
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Michiel Kuijpers (Other)
Responsible Party: Sponsor-Investigator, Michiel Kuijpers, MD, University of Groningen
Organization: University of Groningen (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NL5234.042.15
Record Dates: First submitted 2015-08-25; First posted 2016-02-11 (Estimated); Last update posted 2019-03-04 (Actual); Status verified 2019-02

CONDITIONS: Raynauds

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- All (Experimental): All patient will undergo a unilateral sympathicotomy R3. After this left and right will be compared
  Interventions: Procedure: Sympathicotomy R3

INTERVENTIONS:
Procedure: Sympathicotomy R3 — sympathicotomy R3 consists of transecting the sympathetic chain at the third costal level, cranial of the ganglia, leaving the ganglia themselves untouched

SUMMARY:
The goal is to investigate the effect of a single-port R3 sympathicotomy on microvascular circulation in the affected fingers. This effect is analysed by performing cooling plethysmography and nailfold capillary microscopy bilaterally, following a unilateral, single-port thoracoscopic sympathicotomy.

DETAILED DESCRIPTION:
Raynaud's phenomenon is discoloration, discomfort and numbness or pain in the fingers and toes as a result of excessively reduced blood flow due to sympathetic induced vasospasms, in response to a change in temperature or emotional stress. It usually affects multiple fingers of both hands and comes in frequent attacks, with little or no discomfort in between them. Current treatment consists of stepped-care, including preventive measures optimizing digital blood flow, oral and intravenous medical therapy aimed at improving microvascular circulation, surgical neuromodulation to achieve vasodilatation and neurostimulation.

While surgical sympathectomy is an established treatment of Raynaud's phenomenon, its more invasive nature has prevented widespread application as an initial therapy. After introduction of minimally invasive surgical techniques in recent years, the investigators have further optimized the endoscopic sympathicotomy procedure performed on hyperhidrosis patients, now needing only a single 1 cm port for a detailed, panoramic view of the sympathetic chain (1). This minimal invasive technique has proven to be a safe, efficient and reproducible treatment for several indications and seems also suitable for Raynaud's patients.

In this feasibility study, the researchers want to investigate the effect of a single-port R3 sympathicotomy on microvascular circulation in the affected fingers. This effect is analysed by performing cooling plethysmography and nailfold capillary microscopy bilaterally, following a unilateral, single-port thoracoscopic sympathicotomy.

ELIGIBILITY:
Inclusion Criteria:

* Severe form of SRP, defined as clinical need of prostacyclin analogue infusions and/or bosentan having been given in the preceding 2 years, without satisfying result.
* No concurrent neurological disease

Exclusion Criteria:

* Known Chronic Obstructive Pulmonary Disease > Gold class 1.
* History of smoking > 20 pack years, due to higher risk of complications following unilateral lung- deflation and re-insufflation.
* Documented substance addiction.
* Signs/symptoms of macrovascular disease, or abnormalities on Doppler/duplex studies
* Other signs/symptoms of systemic autoimmune disease
* Severe concomitant diseases of the liver (eg Liver Function tests > three times the upper limit of normal), kidneys (creatinine > 160 mol/l), heart (including history of myocardial infarction, heart failure or angina pectoris), lung, blood, endocrine system, gastrointestinal system, Central Nervous System.
* Previous intra-thoracic pleural drainage.
* Previous thoracic surgery (including sternotomy).
* Gross pulmonary or pleural abnormalities on chest X-ray.
* Pregnancy.
* Unsuitable anatomy (e.g. due to severe physical malformations).

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 8 (Actual)
Dates: Start 2016-02; Primary Completion 2019-02-01 (Actual); Study Completion 2019-02-01 (Actual)

PRIMARY OUTCOMES:
Cooling plethysmography, nailfold capillary microscopy | 1 month follow up
  Change from baseline in microvascular circulation at 1 month
Cooling plethysmography, nailfold capillary microscopy | 6 month follow up
  Change from baseline in microvascular circulation at 6 months

SECONDARY OUTCOMES:
Quality of Life | 1, 6 and 12 months of follow-up
  Change from baseline in quality of life as measured by Short Form 36 (SF36) at 1, 6 and 12 months

CONTACTS AND LOCATIONS:
Locations (1):
- University Medical Centre Groningen, Groningen, Netherlands

REFERENCES:
- [Derived] Kuijpers M, van de Zande SC, van Roon AM, van Roon AM, Stel AJ, Smit AJ, Bouma W, DeJongste MJL, Mariani MA, Klinkenberg TJ, Mulder DJ. Treatment of resistant Raynaud's phenomenon with single-port thoracoscopic sympathicotomy: One-year follow-up. Semin Arthritis Rheum. 2022 Oct;56:152065. doi: 10.1016/j.semarthrit.2022.152065. Epub 2022 Jul 9. PMID 35944349
- [Derived] van Roon AM, Kuijpers M, van de Zande SC, Abdulle AE, van Roon AM, Bos R, Bouma W, Klinkenberg TJ, Bootsma H, DeJongste MJL, Mariani MA, Smit AJ, Mulder DJ. Treatment of resistant Raynaud's phenomenon with single-port thoracoscopic sympathicotomy: a novel minimally invasive endoscopic technique. Rheumatology (Oxford). 2020 May 1;59(5):1021-1025. doi: 10.1093/rheumatology/kez386. PMID 31529103